CLINICAL TRIAL: NCT01407211
Title: The Impact of Vitamin A Supplementation on Gene Expression of Cytokine Secreted by CD4+ T Lymphocyte in Multiple Sclerosis Patients
Brief Title: Impact of Vitamin A on Gene Expression, in Multiple Sclerosis Patient
Acronym: MS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 89/8/18-10033
Record Dates: First submitted 2011-02-14; First posted 2011-08-02 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: multiple sclerosis; Myelin Oligodendrocyte Glycoprotein(MOG); Vitamin A; CD4-Positive T-Lymphocytes; gene expression; Th1 Cells; Th2 Cells
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- with Multiple Sclerosis/ vitamin A (Active Comparator): Patients with Multiple Sclerosis confirmed Relapsing Remitting Type who receive 25000 IU/day vitamin A
  Interventions: Dietary Supplement: vitamin A
- with Multiple Sclerosis/ placebo (Placebo Comparator): Patients with Multiple Sclerosis confirmed Relapsing Remitting Type who receive 1 cap of placebo/day
  Interventions: Dietary Supplement: vitamin A

INTERVENTIONS:
Dietary Supplement: vitamin A — 25000 IU/day vitamin A 6 months
  1 Cap/Day
  1 cap placebo/day for 6 month

SUMMARY:
The aim of this study is the comparison between the effects of supplementation with vitamin A (retinyl palmitate) or placebo for 6 months on gene expression of T CD4+ lymphocyte in multiple sclerotic patient.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic inflammatory demyelinating disease of the central nervous system (CNS).The most important reason for the limited success obtained in the treatment and prevention so far is most likely related to the limited knowledge about its cause and pathogenesis of MS.One of the recent proposed mechanism for autoimmunity base of MS is Th1/Th2 implance of as well as other inflammatory and anti-inflammatory T cell such as Th17 and Treg and their releasing cytokines. Therefore the control of cytokine production may become potential therapeutic targets and modulation of the Th1/Th2 balance may provide a new pharmacological tool to treat this disease. Vitamin A (VA) or VA-like analogs known as retinoids, are potent hormonal modifiers of type 1 or type 2 responses but a definitive description of their mechanism(s) of action is lacking. high level dietary vitamin A enhances Th2 cytokine production and IgA responses, and is likely to decrease Th1 cytokine production. Retinoic acid inhibits IL 12 production in activated macrophages, and RA pretreatment of macrophages reduces IFNγ production and increases IL4 production in antigen primed CD4 T cells. Supplemental treatment with vitamin A or retinoic acid (RA) decreases IFNγ and increases IL5, IL10, and IL4 production. Thus, vitamin A deficiency biases the immune response in a Th1 direction, whereas high level dietary vitamin A may bias the response in a Th2 direction.

ELIGIBILITY:
Inclusion Criteria:

Patients who have used interferon beta in last 3 months. Patients with 1-5 EDSS

Exclusion Criteria:

* Patients who have diseases which affect on Th1/Th2 balance such as asthma, active viral infections, and autoimmune diseases, OR
* Patients who have allergy to vitamin A compounds, OR
* Patients who have used vitamin supplements in last 3 months. -

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
serum Total cholesterol | Change from baseline at 6 months
serum HDL cholesterol | Change from baseline at 6 months
serum triglycerides level | Change from baseline at 6 months
RBP/ TTR ratio | Change from baseline at 6 months
PBMC's prolifration(BrdU colorimetric) | Change from baseline at 6 months
complete blood count (CBC) | Change from baseline at 6 months
serum SGOT concentration | Change from baseline at 6 months
serum SGPT concentration | Change from baseline at 6 months

SECONDARY OUTCOMES:
gene expression of T-bet, INF-gamma, IL-4, GATA3, IL-17, RORc, IL-10, FOXP3 (Relative quantification) | Change from baseline at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran University of Medical Sciences, School of Public Health, Tehran, Iran